CLINICAL TRIAL: NCT02576899
Title: Improving Functional Outcomes of Veterans With PTSD and Tobacco Dependence
Acronym: ACT-PT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1756-P; 121RX-001756-01A1 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2015-10-06; First posted 2015-10-15 (Estimated); Results first posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-03

CONDITIONS: Tobacco; Posttraumatic Stress Disorder
Keywords: smoking cessation; posttraumatic stress disorder; tobacco; treatment; smoking; mindfulness; acceptance; functioning
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Smoking Cessation; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage 1b Study of ACT-PT vs. FFS (Active Comparator): This study involves a randomized clinical trial study of Veteran smokers with PTSD and tobacco dependence randomized to one of two different types of psychosocial treatment: ACT-PT versus the American Lung Association's Freedom From Smoking Program [FFS]. This study has two primary aims: 1) Evaluate the relative feasibility and acceptability of the two interventions (including ease of recruitment, randomization proportion, staff and Veteran acceptance of the treatment, retention rates, treatment adherence, fidelity, ease of the assessment process), and 2) Evaluate the preliminary efficacy of ACT-PT vs. FFS with the primary outcomes of tobacco use, PTSD symptoms, health-related quality of life, and functional impairment.
  Interventions: Behavioral: Acceptance and Commitment Therapy for PTSD and Tobacco Use
- Freedom From Smoking (Placebo Comparator): The American Lung Association's Freedom from Smoking program (FFS) is a commonly used smoking cessation intervention that is used in community treatment programs.
  Interventions: Behavioral: Freedom From Smoking

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy for PTSD and Tobacco Use — ACT-PT is an acceptance and mindfulness-based smoking cessation treatment for Veterans with PTSD and tobacco dependence. ACT-PT specifically targets smoking cravings related to PTSD symptoms and memories of trauma, in addition to difficulties managing PTSD symptoms. negative affect and nicotine withdrawal symptoms during quit attempts. ACT-PT includes structured intervention components that guide Veterans to replace smoking as a coping strategy for PTSD symptoms and memories with alternative coping strategies (e.g., mindfulness, acceptance). And healthy living activities (e.g., engaging in work, expanding social networks, engaging in physical exercise) that are consistent with Veterans' values.
  Arms: Stage 1b Study of ACT-PT vs. FFS
Behavioral: Freedom From Smoking — The American Lung Association's Freedom from Smoking program (FFS) is a commonly used smoking cessation intervention that is used in community treatment programs.
  Arms: Freedom From Smoking

SUMMARY:
Veterans with PTSD have high rates of smoking (34%-86% vs. 18% in the general population) and have substantial difficulties with quitting tobacco. Despite the significant morbidity and mortality associated with smoking, no smoking cessation treatments exist that intensively target PTSD symptoms as an obstacle to quit smoking, although this is a significant barrier to quitting for many Veterans. In addition, no smoking cessation treatments have a large emphasis on improving the functioning of Veterans with PTSD and tobacco dependence, although both PTSD and tobacco use negatively affect functioning across physical, mental health, and social domains.

The goal of this SPiRE project is to evaluate Acceptance and Commitment Therapy for Veterans with PTSD and Tobacco Use (ACT-PT), which is an acceptance and mindfulness-based smoking cessation treatment for Veterans with PTSD and tobacco dependence. ACT-PT specifically targets smoking cravings related to PTSD symptoms and memories of trauma, in addition to difficulties managing PTSD symptoms. negative affect and nicotine withdrawal symptoms during quit attempts. ACT-PT includes structured intervention components that guide Veterans to replace smoking as a coping strategy for PTSD symptoms and memories with alternative coping strategies (e.g., mindfulness, acceptance). And healthy living activities (e.g., engaging in work, expanding social networks, engaging in physical exercise) that are consistent with Veterans' values.

This project involves a small randomized clinical trial study of Veteran smokers with PTSD and tobacco dependence randomized to one of two different types of psychosocial treatment: ACT-PT versus the American Lung Association's Freedom From Smoking Program [FFS]. This study has two primary aims: 1) evaluate the relative feasibility and acceptability of the two interventions (including ease of recruitment, randomization proportion, staff and Veteran acceptance of the treatment, retention rates, treatment adherence, fidelity, ease of the assessment process), and 2) evaluate the preliminary efficacy of ACT-PT vs. FFS with the primary outcomes of tobacco use, PTSD symptoms, health-related quality of life, and functional impairment.

DETAILED DESCRIPTION:
Veterans with PTSD have high rates of smoking (34%-86% vs. 18% in the general population) and have substantial difficulties with quitting tobacco. Only 23% of individuals with PTSD quit smoking compared to 50% of the general population. As a result, Veterans with PTSD are at high risk of developing severe health problems and poor physical functioning. Fifty percent of these long-term smokers will die of a smoking-related cause and on average, will lose 25 years of their life compared to non-smokers. Despite the significant morbidity and mortality associated with smoking, no smoking cessation treatments exist that intensively target PTSD symptoms as an obstacle to quit smoking, although this is a significant barrier to quitting for many Veterans. In addition, no smoking cessation treatments have a large emphasis on improving the functioning of Veterans with PTSD and tobacco dependence, although both PTSD and tobacco use negatively affect functioning across physical, mental health, and social domains.

The goal of this SPiRE project is to evaluate Acceptance and Commitment Therapy for Veterans with PTSD and Tobacco Use (ACT-PT), which is an acceptance and mindfulness-based smoking cessation treatment for Veterans with PTSD and tobacco dependence. ACT-PT specifically targets smoking cravings related to PTSD symptoms and memories of trauma, in addition to difficulties managing PTSD symptoms. negative affect and nicotine withdrawal symptoms during quit attempts. ACT-PT includes structured intervention components that guide Veterans to replace smoking as a coping strategy for PTSD symptoms and memories with alternative coping strategies (e.g., mindfulness, acceptance). And healthy living activities (e.g., engaging in work, expanding social networks, engaging in physical exercise) that are consistent with Veterans' values. This emphasis on substantially improving health-related quality of life and functioning across several areas makes ACT-PT particularly innovative and different from existing treatments. However, research is needed on the relative feasibility, acceptability, and efficacy of ACT-PT compared to standard smoking cessation treatments.

This project involves a randomized clinical trial study of Veteran smokers with PTSD and tobacco dependence randomized to one of two different types of psychosocial treatment: ACT-PT versus the American Lung Association's Freedom From Smoking Program [FFS] with all participants. This study has two primary aims: 1) evaluate the relative feasibility and acceptability of the two interventions (including ease of recruitment, randomization proportion, staff and Veteran acceptance of the treatment, retention rates, treatment adherence, fidelity, ease of the assessment process), and 2) evaluate the preliminary efficacy of ACT-PT vs. FFS with the primary outcomes of tobacco use, PTSD symptoms, health-related quality of life, and functional impairment.

ELIGIBILITY:
Inclusion Criteria:

* Veterans enrolled at the Edith Nourse Rogers Memorial Veterans Hospital
* Current Diagnostic and Statistical Manual (DSM-5) Diagnosis of PTSD
* Minimum score of 38 (clinical cutoff for PTSD) on the PTSD Checklist for DSM-5
* A regular smoker for at least 3 years
* Currently smoking at least 10 cigarettes per day
* Able to communicate meaningfully with the investigator
* Competent to provide written informed consent
* Ages 18 and older

Exclusion Criteria:

* Current unstable DSM-5 bipolar disorder [i.e., instability characterized by two or more manic or depressive episodes in the past 12 months, and a current Young Mania Rating Scale total score of 13 or a current Beck Depression Inventory (BDI) score of 19]
* Any lifetime DSM-5 psychotic disorder
* Current or recent (within 1 month of study entry) moderate or severe DSM-5 alcohol or drug use disorder
* Use of other tobacco products
* A cognitive impairment that would interfere with participation
* A suicide attempt or severe suicidal ideation within the past 3 months
* Presence of any clinical features requiring inpatient or partial hospital treatment
* Use of any other tobacco cessation counseling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan M Kelly, PhD MS, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1b Study of ACT-PT vs. FFS: This study involves a randomized clinical trial study of 50 Veteran smokers with PTSD and tobacco dependence randomized to one of two different types of psychosocial treatment: 10 individual sessions of ACT-PT (n= 25) versus 10 individual sessions of the American Lung Association's Freedom From Smoking Program [FFS] (n=25). This study has two primary aims: 1) Evaluate the relative feasibility and acceptability of the two interventions (including ease of recruitment, randomization proportion, staff and Veteran acceptance of the treatment, retention rates, treatment adherence, fidelity, ease of the assessment process), and 2) Evaluate the preliminary efficacy of ACT-PT vs. FFS with the primary outcomes of tobacco use, PTSD symptoms, health-related quality of life, and functional impairment.
  Acceptance and Commitment Therapy for PTSD and Tobacco Use: ACT-PT is an acceptance and mindfulness-based smoking cessation treatment for Veterans with PTSD and tobacco dependence.
Period: Overall Study
Arm/Group | Stage 1b Study of ACT-PT vs. FFS | Freedom From Smoking
Started | 16 | 20
Completed | 5 | 7
Not Completed | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- ACT-PT: Acceptance and Commitment Therapy for PTSD and Tobacco Use: ACT-PT is an acceptance and mindfulness-based smoking cessation treatment for Veterans with PTSD and tobacco dependence.
- Total: Total of all reporting groups
Arm/Group | ACT-PT | Freedom From Smoking | Total
Number analyzed (Participants) | 16 | 20 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.7 (12.3) | 52.6 (12.9) | 50.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 13 | 16 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 19 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 19 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 20 | 36
Number of Cigarettes [Mean (Standard Deviation); unit: Number of cigarettes smoked] | 21.1 (10.0) | 24.3 (7.5) | 22.5 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence of Smoking Abstinence
Description: Smoking outcomes will include a self-report of the number of cigarettes smoked at end of treatment, 1-month follow-up, and the 3-month follow-up, verified by carbon monoxide (CO) breath tests (< 8 ppm).
Time Frame: Change in smoking abstinence from Baseline to End of Treatment (12 week outcome)
Measure: Count of Participants; unit: Participants
Arm/Group | ACT-PT | Freedom From Smoking
Number analyzed (Participants) | 16 | 20
Participants | 4 | 0

2. Primary Outcome: PTSD Symptoms as Measured by the PTSD Checklist (PCL-5)
Description: The PCL-5 is a brief, self-report symptom checklist that assesses the 20 symptoms of PTSD outlined in the Diagnostic and Statistical Manual-5 (DSM-5) and was designed to assess symptom changes during and after treatment in addition to screening. The PCL has shown satisfactory temporal stability, internal consistency, test-retest reliability, and convergent validity. The minimum value of the PCL-5 is 0, and the maximum value is 80. Higher scores indicate more severe PTSD symptoms.
Time Frame: Change in PTSD symptoms from Baseline to End of Treatment (12 week outcome)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT-PT | Freedom From Smoking
Number analyzed (Participants) | 16 | 20
units on a scale | 38.8 (16.9) | 44.6 (19.2)

3. Primary Outcome: Functional Impairment as Measured by the Mental Health Subscale of The Short Form 36 Health Survey (SF-36)
Description: The Short Form 36 Health Survey (SF-36) is a 36-item self-report measure of current physical, mental health, and social functioning. We are reporting the mental health functioning outcome. A total score was computed by summing and transforming the five-item scores into a score between 0 (lowest mental health) and 100 (highest mental health). Lower scores indicate more severe functioning related to mental health problems.
Time Frame: Change in Functional Impairment from Baseline to End of Treatment (12 week outcome)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ACT-PT: Acceptance and Commitment Therapy for PTSD and Tobacco Use: ACT-PT is an acceptance and mindfulness-based smoking cessation treatment for Veterans with PTSD and tobacco dependence. ACT-PT specifically targets smoking cravings related to PTSD symptoms and memories of trauma, in addition to difficulties managing PTSD symptoms. negative affect and nicotine withdrawal symptoms during quit attempts. ACT-PT includes structured intervention components that guide Veterans to replace smoking as a coping strategy for PTSD symptoms and memories with alternative coping strategies (e.g., mindfulness, acceptance). And healthy living activities (e.g., engaging in work, expanding social networks, engaging in physical exercise) that are consistent with Veterans' values.
Arm/Group | ACT-PT | Freedom From Smoking
Number analyzed (Participants) | 16 | 20
units on a scale | 51.3 (17.8) | 44.3 (21.0)

4. Primary Outcome: Quality of Life as Measured by the Quality of Life Enjoyment and Satisfaction Questionnaire
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire is a commonly used self-report measure to assess quality of life in several domains: general activities, physical health, subjective feelings, leisure time activities, social relationships, work, and household duties. Higher scores indicate better enjoyment and satisfaction with life. The scoring of the Quality of Life Enjoyment and Satisfaction Questionnaire involves summing the first 14 items to yield a total score. The total score ranges from 14 to 70 and is expressed as a percentage based on the maximum total score of the items completed (0-100).
Time Frame: Change in Quality of Life from Baseline to from Baseline to End of Treatment (12 week outcome)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT-PT | Freedom From Smoking
Number analyzed (Participants) | 15 | 19
units on a scale | 44.3 (11.5) | 37.5 (6.3)

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | ACT-PT | Freedom From Smoking
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/20
Other Adverse Events (participants affected / at risk) | 0/16 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT02576899/Prot_SAP_000.pdf